CLINICAL TRIAL: NCT05690919
Title: A Study Analyzing Brain Injury Patients Experience Patterns in Medical Trials
Brief Title: Examining the Experiences of Brain Injury Patients in Medical Trials
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 84028751
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Brain Injuries
Keywords: Brain Injuries
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Historically, participation in clinical trials has been skewed towards certain groups. However, research on the factors that influence participation, both positive and negative, is limited.

Brain injury clinical trial patients help us identify these factors by sharing trial experiences during the course of the interventional medical study.

This study will include a diverse group of participants to gather a wide range of information on clinical trial experiences. The collected data will then be used to benefit future brain injury patients who are considering participating in a medical study.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with brain injury
* Patient is 18 years old
* Patient has self-identified as planning to enroll in an interventional clinical trial

Exclusion Criteria:

* Patient does not understand, sign, and return consent form
* Patient is pregnant
* Inability to perform regular electronic reporting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Brain injury patients who are actively considering enrolling in an intensive clinical trial, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to enroll in a brain injury clinical trial. | 3 months
Rate of patients who remain in brain injury clinical trial to trial completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Maas AI, Roozenbeek B, Manley GT. Clinical trials in traumatic brain injury: past experience and current developments. Neurotherapeutics. 2010 Jan;7(1):115-26. doi: 10.1016/j.nurt.2009.10.022. PMID 20129503
- [Background] Wat R, Mammi M, Paredes J, Haines J, Alasmari M, Liew A, Lu VM, Arnaout O, Smith TR, Gormley WB, Aglio LS, Mekary RA, Zaidi H. The Effectiveness of Antiepileptic Medications as Prophylaxis of Early Seizure in Patients with Traumatic Brain Injury Compared with Placebo or No Treatment: A Systematic Review and Meta-Analysis. World Neurosurg. 2019 Feb;122:433-440. doi: 10.1016/j.wneu.2018.11.076. Epub 2018 Nov 20. PMID 30465951
- [Background] Kjeldsen SS, Brodal L, Brunner I. Activity and rest in patients with severe acquired brain injury: an observational study. Disabil Rehabil. 2022 Jun;44(12):2744-2751. doi: 10.1080/09638288.2020.1844317. Epub 2020 Nov 8. PMID 33161752

DOCUMENTS (1):
  • Informed Consent Form (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/19/NCT05690919/ICF_000.pdf